CLINICAL TRIAL: NCT06825026
Title: Observatory of the Older Person: A Cohort of Older Adults Living in Nursing Homes in Porto Metropolitan Area
Brief Title: Observatory of the Older Person: A Cohort of Older Adults Living in Nursing Homes
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Maria Joana Carvalho, Principal Investigator, Universidade do Porto
Other Study IDs: CEFADE012021_B
Record Dates: First submitted 2025-01-30; First posted 2025-02-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Frailty
Keywords: Frail; Nursing homes
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pragmatic exercise trial — As part of the broader Observatory of the Older Person cohort, we aim to conduct a pragmatic exercise trial in a subgroup of nursing home residents. This trial seeks to evaluate the effectiveness of a concurrent exercise intervention on frailty, functional capacity, independence in activities of daily living and falls rate in real-world settings.

SUMMARY:
This cohort of older adults residing in nursing homes in Porto Metropolitan Area aims to monitor the health, intrinsic capacity and functional capacity over time. Through systematic data collection and analysis, the observatory provides valuable insights into aging, frailty, and long-term care needs, informing policies and interventions to enhance older adults care. This cohort aims to recruit 400 individuals aged 65 years or more at baseline.All participants will be invited for a re-assessment every year, while the overall duration is planned for four years.

DETAILED DESCRIPTION:
The Observatory of the Older Person is a cohort study designed to enhance understanding of the aging process among older adults in nursing homes. The study aims to generate insights into the determinants of functional and intrinsic capacity, identify factors influencing independence, and develop targeted interventions to improve well-being in this population.

Specifically, it aims:

* To provide a comprehensive characterization of the health profiles across nursing home population. This will include demographic, clinical, and functional assessments, as well as an exploration of variations in health conditions, nutritional status, cognitive function, and psychosocial well-being among residents.
* to examine the trajectories of functional and intrinsic capacity over time by tracking changes in mobility, strength, balance, cognitive function, psychological resilience, and physiological health.
* To determine the key factors contributing to the loss of independence in basic activities of daily living (ADLs). Physical, cognitive, psychological, and social determinants will be analyzed to identify their role in maintaining or reducing autonomy among nursing home residents.
* To investigate the risk factors associated with falls in nursing home residents. Physical frailty, cognitive impairment, polypharmacy, and environmental hazards will be examined to determine their contribution to fall risk. Additionally, the consequences of falls, including injuries, hospitalizations, and fear of falling, will be assessed to evaluated.
* To implement and assess the impact of exercise interventions designed to mitigate or reverse frailty. Tailored programs focusing on strength and endurance will be evaluated for their effectiveness in improving frailty status, reducing fall risk, and promoting autonomy among older adults.

By addressing these objectives, this study will contribute to evidence-based strategies for improving health, independence, and quality of life in nursing home residents.All participants will be invited for a re-assessment every year, while the overall duration is planned for four years. Findings may also inform policies and best practices to enhance care models within long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 or older

Exclusion Criteria:

* Any contraindication that could affect physical exercise performance or testing procedures, including terminal illness, uncontrolled disease, or other unstable medical condition;
* bone fracture in the past 3 months;
* Iinability to understand and follow the instructions of physical tests

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals living in public nursing homes in Porto Metropolitan Area
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
short physical performance battery (SPPB) | 4 years
  The Short Physical Performance Battery (SPPB) is a standardised assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).

SECONDARY OUTCOMES:
Handgrip strength | 4 years
  Handgrip strength will be obtained with a Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA).Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 15s between trials
Barthel Index | 4 years
  The Barthel Index (BI) is a standardized tool used to assess a person's ability to perform activities of daily living (ADLs) independently. It measures 10 basic functions, including feeding, bathing, dressing, toileting, mobility, and stair climbing, with scores ranging from 0 (fully dependent) to 100 (fully independent)
Falls in the last 12 months | 4 years
  A retrospective review of electronic medical records (EMRs) to identify and document instances of falls reported within the last 12 months
Falls rate | 4 years
  A retrospective review of electronic medical records (EMRs) to identify athe number of falls reported within the last 12 months
Frailty status | 4 years
  The frailty phenotype is a clinical model that identifies frailty in older adults based on five criteria: unintentional weight loss, exhaustion, low physical activity, slow walking speed, and weak grip strength. Individuals meeting three or more criteria are classified as frail, two as pre-frail, and none as robust. It helps in identifying at-risk individuals for adverse outcomes and targeting interventions to prevent further decline.

OTHER OUTCOMES:
Times Using the Healthcare System in the Last 6 Months | 4 years
  The number of healthcare encounters (e.g., hospital admissions, emergency department visits, outpatient consultations, and telehealth appointments) within the past six months
Mini Mental State Examination | 4 years
  The Mini-Mental State Examination (MMSE) is a brief, structured tool used to assess cognitive function and screen for dementia. It consists of 30 questions covering areas such as orientation, memory, attention, language, and visuospatial skills. The MMSE is scored out of 30, with higher scores indicating better cognitive function. It is widely used in clinical settings to detect cognitive impairments, monitor changes in cognitive function over time, and assess the severity of cognitive decline. Scores are interpreted based on age and education level, with a lower score suggesting potential cognitive deficits.
Mini Nutritional Assessment Short Form (MNA-SF) | 4 years
  The Mini Nutritional Assessment Short Form (MNA-SF) is a simplified version of the Mini Nutritional Assessment (MNA) designed to quickly assess the nutritional status of older adults. It consists of 6 questions, covering aspects such as weight loss, mobility, and food intake, which provide a quick screening for malnutrition risk. The MNA-SF is useful for identifying individuals who may be at risk of malnutrition and is often used in clinical settings for routine assessments. Based on the score, individuals are categorized as well-nourished, at risk of malnutrition, or malnourished, allowing for timely nutrition interventions.
Weight | 4 years
  Assessment of body weight using Inbody 120, which is a body composition analyzer that uses bioelectrical impedance analysis (BIA).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Joana Carvalho, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Sports, University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No